CLINICAL TRIAL: NCT05467904
Title: A Double-Blind Randomized, Placebo-Controlled Trial of a Proprietary Full Hemp Flower Formulation ( Xltran™ and Xltranplus™) to Determine Clinical Improvement in the Syndrome of Long COVID
Brief Title: Double-Blind Randomized Placebo-Controlled Trial of a Proprietary Full Hemp Flower Formulation for Long COVID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: LUCINDA BATEMAN, MD (Other)
Collaborators: Endourage, LLC (Industry)
Responsible Party: Sponsor-Investigator, LUCINDA BATEMAN, MD, Medical Director, Bateman Horne Center
Organization: Bateman Horne Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: BHC402-2022
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-03

CONDITIONS: Post-acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Xltranplus (Active Comparator): Xltanplus is a full hemp flower formulation with cannabinoids and terpenes
  Interventions: Other: Xltranplus, Xltran
- Xltran (Active Comparator): Xltran contains terpenes extracted from the hemp flower
  Interventions: Other: Xltranplus, Xltran
- Placebo (Placebo Comparator): Placebo will be an inactive formulation of water, sunflower lecithin and polysorbate
  Interventions: Other: Xltranplus, Xltran

INTERVENTIONS:
Other: Xltranplus, Xltran — Xltranplus and Xltran are full hemp flower formulations

SUMMARY:
This is a double-blind, randomized, placebo-controlled single-center clinical trial to explore the safety and efficacy of a full cannabis flower formulation, rich in cannabinoids and terpenes formulation, Xltran Plus™ and Xltran™, both compared to placebo for the treatment of Long COVID patients with prolonged symptoms caused by COVID-19.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled single-center, 28-day study designed to explore the safety and efficacy of Xltran Plus™ and Xltran™ for the treatment of Long COVID in adults. The treatment consists of daily doses of Xltran Plus™, Xltran™, or placebo. Xltran Plus™ contains 10.42 mg of cannabinoids, 0.55 mg tetrahydrocannabinol (THC), and 2.729 mg of terpenes per 0.25 ml of solution. Xltran™ contains 0 mg of cannabinoids, 0 mg THC and 1.28 mg terpene per 0.25 ml of solution. Placebo contains water, sunflower lecithin and polysorbate. Trial participants will be randomized to Xltran Plus™, Xltran™ or placebo at Visit 1. Participants will take 1 ml sublingually after morning meal and 1 ml sublingually after the evening meal for 28 days.

There will be 111 patients with Long COVID enrolled. There will be approximately 37 patients randomized to each arm.

Candidates will undergo initial pre-screening by telephone, after which, if they appear to meet initial entry criteria, will be invited for an in-person visit. The first visit, Visit 1, will include vitals, symptom questionnaires, cognitive testing, and urine and blood sampling. Participants will receive weekly symptom surveys to complete online. Each participant will be instructed on cognitive testing using their smart phone and complete the cognitive testing weekly.

Patients with underlying medical or psychiatric conditions that could impact their safe participation in the study or interfere with their ability to complete or comply with the study's requirements will not be enrolled. Patients on active illicit or non-prescribed drug use and chronic, daily use of an immune suppressant (e.g., prednisone) will be excluded. Patients with documented history and active treatment for seizure disorder, and any condition that in the opinion of the investigator would be harmful or detrimental to the patient will not be enrolled in the study.

Patients may remain on stable doses of opioids, SSRIs and other anti-depressants; however, poorly controlled, or severely depressed patients will not be enrolled. Only clinically stable and well-controlled patients will be considered.

At Visit 1, the PI will ensure that all entry criteria have been satisfied and the participant will be randomized and initiate treatment with one dose on the day of the Visit 1 (Day 1), followed by BID dosing for the duration of the study.

Urine will be collected at Visit 1 for pregnancy testing. Urine drug screening for drugs of abuse will be conducted at Visit 1; patients positive for cocaine, methamphetamine, phencyclidine (PCP), methadone, non-disclosed opiates, or marijuana metabolites should be screen failed. Patients positive for disclosed, stable doses of prescribed opioids are able and may remain on these medications during the study. Additional drug testing may be conducted at the investigator's discretion.

A blood sample will be collected at Day 1 (Visit 1) and Day 28 (Visit 2) for changes in inflammatory markers.

Patients will receive assigned study treatment for a total of 28 days, with treatment dispensed at Visit 1 (Day 1) and the amount of treatment remaining, if any, accounted for at Visit 2 (Day 28) end of treatment visit.

At the end of the trial and after results are unblinded, those who received placebo will be provided with a 28-day supply each of Xltran Plus™ and Xltran™ if they are interested.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to read, understand, and sign the informed consent
2. Diagnosis of Long COVID is defined as the following:

   1. Infected individuals will have a confirmed SARS-CoV-2 infection within 36 months of enrollment and have had at least one month of persistent fatigue and muscle weakness, functional impairment, and cognitive impairment since the acute infection.
   2. Adults with confirmed prior SARS-CoV-2 infection will satisfy any one of the following:

   i. Any person with a positive SARS-CoV-2 polymerase chain reaction (PCR) or nucleic acid amplification test (NAAT); ii. Any person with a positive SARS-CoV-2 antigen rapid diagnostic test; iii. Any person with a positive SARS-CoV-2 antibody test
3. Male and female patients, 18-65 years of age

   a. Female patients of child-bearing potential must have a negative urine pregnancy test at Visit 1. Women confirmed to be of non-childbearing potential do not require pregnancy testing. To be considered of non-child-bearing potential, the patient must be: i. Post-menopausal (defined as no menses for at least one year); or ii. Surgically sterile (s/p hysterectomy, bilateral oophorectomy, or bilateral tubal ligation at least six months prior to beginning treatment with study product); or iii. At least three months s/p a non-surgical permanent sterilization procedure b. Females of child-bearing potential must be willing to utilize an effective birth control method for the duration of the study. Women involved in monogamous same-sex relationships or committed to sexual abstinence (e.g., religious reasons) will be waived from this requirement. Allowable contraceptive methods include: i. Oral, implantable, injectable, or transdermal hormonal contraceptives (should have been used for a minimum of one full cycle prior to administration of study product) ii. Intrauterine devices (IUD) iii. Vasectomized partner iv. Double barrier method (male or female condom, sponge, diaphragm, or vaginal ring with simultaneous use of spermicidal jelly or cream)
4. A urine drug screen performed at the Visit 1 must be negative for drugs of abuse such as methamphetamine, cocaine, phencyclidine (PCP), marijuana metabolites, and non-disclosed amphetamines and opioids/opiates. The following stipulations also apply:

   a. Patients with a positive screening UDS due to prescribed amphetamines for allowed conditions do not require further UDS testing. They may proceed with study treatment, assuming no evidence of abuse or dependency.
5. Patients should not require treatment with warfarin, heparin, lithium, digoxin, amiodarone, isoniazid, phenytoin, fluconazole, methotrexate, probenecid, or raloxifene. Patients on these medications should not be screened.
6. Patients agree to refrain from taking medications that would affect assessment of the effectiveness of study product for the duration of the study
7. Willing and able to comply with all protocol-specified requirements
8. Have a smart phone and internet access to complete online surveys and cognitive testing

   Exclusion Criteria:
9. Improvement in fatigue and physical function because of any treatment intervention in the past month
10. Use of Xltran Plus™ or Xltran™ within 30 days of Visit 1.
11. Current use of marijuana or medical cannabis
12. Currently receiving chronic/daily systemic corticosteroids (>5 mg prednisone daily, or equivalent)
13. BMI <20 or >40
14. Breastfeeding or pregnant, or planning to become pregnant during the next six months
15. In the opinion of the Investigator, any clinically significant, uncontrolled, or unstable medical or surgical condition that could affect the patient's ability to participate in the study or potentially compromise their well-being while enrolled in the study

    a. Symptomatic and/or otherwise clinically significant cardiac disease, including but not limited to: myocardial infarction during the preceding two years; uncontrolled hypertension; symptomatic heart failure (e.g., New York Heart Association Class II or higher); angina or other evidence of significant coronary artery disease; or anticipation of bypass or other cardiac surgery within the next 12 months
16. In the opinion of the Investigator, evidence of a clinically significant psychiatric disorder; e.g., severe, unstable or poorly controlled depression, anxiety or obsessive-compulsive disorder; moderate or severe alcohol use disorder; substance use disorder; or any history of bipolar disorder, schizophrenia, schizoaffective disorder or other psychotic disorder
17. History of suicide attempt or other suicidal behavior in the previous two years.
18. Any anticipated need for surgery that might confound results or interfere with the patient's ability to comply with the protocol
19. Known allergies to hemp seeds, medical cannabis, sunflower lecithin or polysorbate
20. Current enrollment in any other research or clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) | Change in PGIC from beginning to end of treatment at 30 days
  PGIC is a 7 point scale rating individuals perception of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Total Symptom Score (TSS) | Change in TSS from beginning to end of treatment at 30 days
  TSS is the sum of patient-reported scores (0-5 scale, 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, and 5=very severe) for each of 10 symptoms, specifically: (i) fatigue/weakness; (ii) pain, e.g., musculoskeletal, allodynia; (iii) brain fog; (iv) dysautonomia, e.g., tachycardia, hypotension, orthostatic intolerance, dizziness, vertigo, light-headedness, syncope, gastrointestinal/urinary issues; (v) headaches, including head/neck discomfort; (vi) sensory problems, e.g., sensitivity to light, sound, odor, taste, touch, or problems such as blurry vision, tinnitus, etc; (vii) sleep difficulties; (viii) shortness of breath; (ix) flu-like symptoms, e.g., sore throat, tender lymph nodes, feverishness, sinus or nasal congestion; and (x) mood disorders, e.g., anxiety, depression.

SECONDARY OUTCOMES:
Insomnia Severity Index | Univariate time series analysis of change/trend of weekly responses over 30 days
  A brief 7 item instrument to assess the severity of both nighttime and daytime components of insomnia
Harvard Flourishing Index (HFI) | Univariate time series analysis of change/trend of weekly responses over 30 days
  Consists of two questions or items from each of the five main subscales: happiness and life satisfaction, mental and physical health, meaning and purpose, character and virtue, and close social relationships.
DANA Brain Vital | Univariate time series analysis of change/trend of weekly cognitive efficiency over 30 days
  Assessment of reaction time cognitive efficiency
Hours of Upright Activity | Univariate time series analysis of change/trend of daily responses over 30 days
  Self-reported time with feet on the floor over a 24 hours period
Daily Steps | Univariate time series analysis of change/trend of daily steps over 30 days
  Daily steps over a 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda Bateman, MD, Principal Investigator — Chief Medical Officer
Locations (1):
- Bateman Horne Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No